CLINICAL TRIAL: NCT01366794
Title: Effects of Macronutrients on Gut Hormone and Islet Hormone Secretion in Healthy Volunteers and Type 2 Diabetes
Brief Title: Macronutrients and Gut Hormone Secretion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Bo Ahren, Professor, Lund University
Allocation: Non-Randomized | Model: Factorial | Masking: None
Other Study IDs: 005
Record Dates: First submitted 2011-05-31; First posted 2011-06-06 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Type 2 Diabetes
Keywords: Gut hormones; Insulin secretion
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Nutrients; Glucose; soybean oil, phospholipid emulsion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Type 2 diabetes (Experimental): Administration of macronutrients in type 2 diabetes
  Interventions: Other: Macronutrients
- Healthy volunteers (Experimental): Administration of macronutrients in healthy volunteers
  Interventions: Other: Macronutrients

INTERVENTIONS:
Other: Macronutrients — Glucose 330 kcal Protein 110 kcal Fat emulsion 110 kcal Mixed meal 550 kcal
  Other Names: Glucose; Protein mixture; Fat emulsion; Mixed meal

SUMMARY:
Study hypothesis is to examine the relative contribution of macronutrients for gut hormone secretion after a mixed meal in healthy volunteers and in subjects with type 2 diabetes. Individual macronutrients or a mixed meal will therefore be served and gut hormones are measured during the following 300 min.

DETAILED DESCRIPTION:
In healthy volunteers and subjects with dietary regulated diabetes mellitus, glucose, protein mixture or fat emulsion will be served individually and on a separate occasions a mixed meal will be served. Samples will be taken during the following 300 min. Concentrations of the gut hormones glucose-dependent insulinotropic polypeptide and glucagon-like peptide-1, insulin and glucagon will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Healthy status or type 2 diabetes with dietary regulation

Exclusion Criteria:

* Liver disease
* kidney disease
* thyroid disease

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Release of gut hormones | 300 min

SECONDARY OUTCOMES:
Insulin secretion | 300 min

CONTACTS AND LOCATIONS:
Overall Officials: Bo Ahrén, PhD, Principal Investigator — Lund University
Locations (2):
- Sweden (2):
  - Department of Clinical Sciences Lund, Lund University, Lund
  - Lund University, Lund